CLINICAL TRIAL: NCT06518252
Title: Detection of the Risk of Sudden Cardiac Death in Athletes From the Universidad Nacional de Colombia
Brief Title: Risk of Sudden Cardiac Death in UN Athletes
Acronym: Suddendeath
Status: Recruiting | Type: Observational
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Other Study IDs: B.FM.1.002-CE-225-23
Record Dates: First submitted 2024-06-12; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Death, Sudden, Cardiac; Electrocardiogram QT Prolonged; Athlete Heart; Athletic Injuries
Keywords: Sudden death of the athlete; Electrocardiogram; University sports.
MeSH Terms: conditions — Death, Sudden, Cardiac; Long QT Syndrome; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The detection of sudden cardiac death risk in athletes is a topic of great relevance in the field of sports physiotherapy and physical activity. High-performance sports practice involves anatomical and physiological changes that can modify the mechanical and electrical properties of the heart, increasing the risk of potentially fatal cardiac events. Therefore, it is essential to implement early detection strategies to identify at-risk athletes and prevent tragedies during sports practice.

Methodology: This study focuses on the prevalence of sudden cardiac death risk, using a 12-lead electrocardiogram as the primary detection tool. This examination will allow for the evaluation of the heart's electrical activity and the detection of potential anomalies that could predispose athletes to adverse cardiac events during sports practice. In addition to the electrocardiogram, cardiovascular screening questionnaires will be administered to collect information on personal and family health histories, as well as other relevant risk factors. In conjunction with the project's researchers, the sports medical team of the Universidad Nacional de Colombia will be responsible for conducting the evaluations, ensuring the precision and reliability of the obtained results. A detailed analysis of the collected data will be performed using statistical tools to identify possible correlations between the evaluated risk factors and the presence of sudden cardiac death risk in athletes. Logistic regression models will be employed to determine the strength of association between the studied variables and cardiovascular risk in this specific population.

Expected Results: It is anticipated that implementing pre-participation evaluations, including the electrocardiogram and cardiovascular screening questionnaires, will enable the identification of athletes at higher risk of sudden cardiac death. These results will allow for the establishment of individualized risk profiles and the design of personalized prevention strategies for each athlete. Additionally, it is expected that the findings of this study will contribute to the development of early detection protocols for sudden cardiac death risk in athletes, which can be effectively implemented in sports settings. The information generated from this study will provide a solid foundation for clinical decision-making and the implementation of preventive measures to benefit the health and well-being of high-performance athletes.

DETAILED DESCRIPTION:
Methodological Framework Research Question: What is the prevalence of sudden death risk and its predisposing factors in athletes belonging to the sports teams of the Univerisdad Nacional de Colombia - Bogotá campus aged between 18 and 35 years?

General Objective: To identify the prevalence of sudden death risk and its predisposing factors in athletes belonging to the sports teams of the National University of Colombia - Bogotá campus aged between 18 and 35 years.

Specific Objectives: 1. Characterize athletes belonging to the sports teams based on 12-lead ECG electrocardiographic activity, 2. Establish predisposing risk factors associated with sudden death in UNAL athletes belonging to the sports teams, 3. Determine the relationship between sudden death risk and predisposing factors related to cardiovascular risk, medical history, and training loads, intensities, and volumes.

Working Hypothesis. H1: Among the evaluated athletes, there will be a prevalence of sudden death risk equal to or greater than that reported in the literature. H0: The prevalence of sudden death risk found in the research will be lower than that reported in the literature.

Statistical Hypothesis. H1: The risk of sudden death is 3% to 5% higher in an athlete compared to a non-athlete. H0: The risk of sudden death is less than 3% in an athlete compared to a non-athlete.

Recruitment and Dissemination of Research Project Call. A recruitment process for participants will be carried out using an internal engagement model targeting members of the UNAL sports teams through the snowball sampling method.

Protocol for ECG Acquisition. The examination to be used for the application of a 12-lead electrocardiogram (ECG) to detect the risk of sudden death in athletes, considered the Gold Standard by the SEC and AHA. There are 6 precordial leads, and 4 limb leads, both upper and lower limbs. The person responsible for the ECG acquisition will be the principal investigator, who has completed the full course on ECG acquisition and interpretation from the Colombian Association of Cardiology and Cardiovascular Surgery. In case the principal investigator cannot participate in the complete acquisition of the ECG, the sports medicine physician from the specific area will perform the acquisition. The following protocol for ECG acquisition will be used:

1. Subject reception.
2. Registration of personal information and sports modality.
3. Review of ECG acquisition criteria.
4. Explanation of the procedure to the athlete (it is crucial to emphasize that they should not move during the examination as this may alter the results).
5. Explanation of the informed consent process (Annex 2), procedures to be performed, potential results, benefits, and assurance of respect and confidentiality of the collected information during the research, followed by signing the informed consent form.
6. A rest period of 2 minutes in complete calmness.
7. Inquiry about and removal of metallic items in the body such as prosthetics, hearing aids, piercings, among others, that may cause interference in the results.
8. Cleaning of the areas where the electrodes will be placed, both central and peripheral. This cleaning can be done with 70% alcohol wipes.
9. Application of conductive gel on each electrode, both central and peripheral.
10. Placement of each electrode in each site: 6 precordial, 2 on upper limbs, and 2 on lower limbs.
11. Recording the electrocardiogram for 2 minutes.
12. After the ECG acquisition, removal of electrodes and excess conductive gel.
13. Delivery of ECG results to the sports medicine specialist, who reads and records the findings of the examination.

In addition to the acquisition, there is also a registration process that must be done when interpreting an ECG: 1. Full name of the patient, 2. Sports discipline, 3. Taking or verifying the heart rate, 4. Determining the presence or absence of risk, 5. Archiving information in folders designated by the researchers.

Statistical Determination Descriptive. For the descriptive analysis of the characteristics of the study population and variables on a qualitative measurement scale, frequencies and proportions will be used. Continuous variables will be described using measures of central tendency (mean and median) and dispersion (standard deviation, interquartile range) according to whether normal distribution is present or not, based on graphical methods (histograms, scatter plots, among others) and numerical methods (Shapiro-Wilk).

Inferential. A correlation analysis will be conducted between secondary variables and their association with sudden death using a logistic regression model. The variables used will include: Age, Gender, Sport modality, Training volume, Training intensity.

Statistics. Prevalence, used to quantify the proportion of individuals in a population at risk of sudden death at the time of measurement, Prevalence rates, quantify the proportion of individuals in a population at risk of sudden death over a certain time, Prevalence difference, used to compare the prevalence described in the research project with that found in other studies with similar methodological characteristics, Odds ratio, used to measure the relationship between athletes exposed to a certain volume and intensity with risk/those who do not present risk.

ELIGIBILITY:
Inclusion Criteria:

* Athletes belonging to the sports teams of the National University of Colombia, Bogotá campus.
* Subject's sports history (practice time exceeding 2 years).
* Individuals aged 18 to 35 years, without discrimination based on biological sex.
* Training time exceeding 6 hours per week in their sports modality (weekly training record).
* Personal history of cardiovascular disease (cardiac malformations or previously detected sudden death risk).
* Athletes who attend at least 90% of the training sessions planned by the coach.

Exclusion Criteria:

* Personal history of metabolic (type 1 and 2 diabetes mellitus), neurological (spinal cord injury), or renal disease.
* Routine consumption of alcohol or psychoactive substances.
* Use of antihypertensive medications, beta-blockers, or inotropes.
* Cardiovascular disease diagnosed with previously established pharmacological management.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Athlete population aged between 18 and 35 years, without excluding gender, belongs to the Universidad Nacional de Colombia (UN), Bogotá campus sports delegations. Measurements will be conducted in the Exercise Physiology Laboratory of the Faculty of Medicine at UN. Se realizará un proceso de reclutamiento de los participantes utilizando un modelo de enganche interno de los pertenecientes a las selecciones deportivas de la UNAL por medio del método bola de nieve.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Sudden death due to ventricular hypertrophy. | 8 months
  People whose electrocardiographic findings are outside the normal parameters and who present left or right ventricular hypertrophy with isolated QRS voltage to the left side (SV1 þ RV5 or RV6 >3.5 mV) or right ventricular hypertrophy (RV1 þ SV5 or SV6 > 1.1mV)
Sudden death due right bundle branch block | 8 months
  People whose electrocardiographic findings are outside normal parameters and presenting rSR0 in V1 and qRS pattern in V6 with QRS duration <120 ms.
Sudden death due to repolarization pattern | 8 months
  People whose electrocardiographic findings are outside the parameters of normality/ST elevation with J point elevation, ST segment elevation, J waves or dragged terminal QRS in the inferior and/or lateral leads
Sudden death due to ST elevation | 8 months
  ST elevation followed by T wave inversion in V1-V4 in black athletes: J-point elevation and convex ("domed") ST segment elevation followed by T wave inversion in leads V1-V4 in athletes black

SECONDARY OUTCOMES:
Sporting modality | 8 months
  Human behavior characterized by a playful and competitive attitude of verification or challenge expressed through physical and mental exercise, within established disciplines and rules. Includes different types of sports according to specific rules and game norms.
Training volume | 8 months
  Training Duration is a quantitative variable that measures the total time spent in an exercise or physical training session. It is expressed in units of time and is understood as the number of minutes of training per week.
Borg scale modified. | 8 months
  Exercise intensity during a training session, measured by coach and athlete self-report using the modified Borg scale with a score from 0 to 10. Scale Description: 0: No effort, 0.5: Very, very light, 1 : Very light, 2: Light, 3: Moderate, 4: Somewhat heavy, 5: Heavy, 6-7: Very heavy, 8-10: Very, very heavy
Weekly Training Frequency | 8 months
  Number of training sessions that a person performs in a week, I understand a training session as the activity planned and carried out for more than 30 minutes. The total number of exercise sessions performed in a week will be taken.

OTHER OUTCOMES:
Age | 8 months
  Time of life that a person has lived since birth. It will include individuals whose ages range from 18 to 35 years old.
Sex | 8 months
  Organic condition that defines individuals as male or female. Individuals will not be discriminated against based on gender.

CONTACTS AND LOCATIONS:
Overall Officials: Wilder Villamil-Parra, PhD.Sciences, Study Director — Universidad Nacional de Colombia; Erica Mancera-Soto, PhD.Sciences, Study Chair — Universidad Nacional de Colombia
Locations (1):
- Juan Murillo-Coca, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han J, Lalario A, Merro E, Sinagra G, Sharma S, Papadakis M, Finocchiaro G. Sudden Cardiac Death in Athletes: Facts and Fallacies. J Cardiovasc Dev Dis. 2023 Feb 5;10(2):68. doi: 10.3390/jcdd10020068. PMID 36826564
- [Background] Sarto P, Zorzi A, Merlo L, Vessella T, Pegoraro C, Giorgiano F, Graziano F, Basso C, Drezner JA, Corrado D. Value of screening for the risk of sudden cardiac death in young competitive athletes. Eur Heart J. 2023 Mar 21;44(12):1084-1092. doi: 10.1093/eurheartj/ehad017. PMID 36760222
- [Background] Sharma S, Drezner JA, Baggish A, Papadakis M, Wilson MG, Prutkin JM, La Gerche A, Ackerman MJ, Borjesson M, Salerno JC, Asif IM, Owens DS, Chung EH, Emery MS, Froelicher VF, Heidbuchel H, Adamuz C, Asplund CA, Cohen G, Harmon KG, Marek JC, Molossi S, Niebauer J, Pelto HF, Perez MV, Riding NR, Saarel T, Schmied CM, Shipon DM, Stein R, Vetter VL, Pelliccia A, Corrado D. International Recommendations for Electrocardiographic Interpretation in Athletes. J Am Coll Cardiol. 2017 Feb 28;69(8):1057-1075. doi: 10.1016/j.jacc.2017.01.015. PMID 28231933
- [Background] Vessella T, Zorzi A, Merlo L, Pegoraro C, Giorgiano F, Trevisanato M, Viel M, Formentini P, Corrado D, Sarto P. The Italian preparticipation evaluation programme: diagnostic yield, rate of disqualification and cost analysis. Br J Sports Med. 2020 Feb;54(4):231-237. doi: 10.1136/bjsports-2018-100293. Epub 2019 Jul 17. PMID 31315826
- [Background] Williams EA, Pelto HF, Toresdahl BG, Prutkin JM, Owens DS, Salerno JC, Harmon KG, Drezner JA. Performance of the American Heart Association ( AHA ) 14-Point Evaluation Versus Electrocardiography for the Cardiovascular Screening of High School Athletes: A Prospective Study. J Am Heart Assoc. 2019 Jul 16;8(14):e012235. doi: 10.1161/JAHA.119.012235. Epub 2019 Jul 9. PMID 31286819
- [Background] Dhutia H, MacLachlan H. Cardiac Screening of Young Athletes: a Practical Approach to Sudden Cardiac Death Prevention. Curr Treat Options Cardiovasc Med. 2018 Aug 28;20(10):85. doi: 10.1007/s11936-018-0681-4. PMID 30155696
- [Background] D'Ascenzi F, Valentini F, Pistoresi S, Frascaro F, Piu P, Cavigli L, Valente S, Focardi M, Cameli M, Bonifazi M, Metra M, Mondillo S. Causes of sudden cardiac death in young athletes and non-athletes: systematic review and meta-analysis: Sudden cardiac death in the young. Trends Cardiovasc Med. 2022 Jul;32(5):299-308. doi: 10.1016/j.tcm.2021.06.001. Epub 2021 Jun 22. PMID 34166791
- [Background] Bassi MD, Farina JM, Bombau J, Fitz Maurice M, Bortman G, Nunez E, Marquez M, Bornancini N, Baranchuk A. Sudden Cardiac Arrest in Basketball and Soccer Stadiums, the Role of Automated External Defibrillators: A Review. For the BELTRAN Study (BaskEtbaLl and soccer sTadiums: Registry on Automatic exterNal defibrillators). Arrhythm Electrophysiol Rev. 2023 Jan;12:e03. doi: 10.15420/aer.2022.30. PMID 36845166
- [Background] Egger F, Scharhag J, Kastner A, Dvorak J, Bohm P, Meyer T. FIFA Sudden Death Registry (FIFA-SDR): a prospective, observational study of sudden death in worldwide football from 2014 to 2018. Br J Sports Med. 2022 Jan;56(2):80-87. doi: 10.1136/bjsports-2020-102368. Epub 2020 Dec 23. PMID 33361135
- [Background] Sims JM. A brief review of the Belmont report. Dimens Crit Care Nurs. 2010 Jul-Aug;29(4):173-4. doi: 10.1097/DCC.0b013e3181de9ec5. PMID 20543620
- [Background] Ehni HJ, Wiesing U. The Declaration of Helsinki in bioethics literature since the last revision in 2013. Bioethics. 2024 May;38(4):335-343. doi: 10.1111/bioe.13270. Epub 2024 Feb 17. PMID 38367022
- [Background] Sweeting J, Semsarian C. Sudden Cardiac Death in Athletes. Heart Lung Circ. 2018 Sep;27(9):1072-1077. doi: 10.1016/j.hlc.2018.03.026. Epub 2018 Apr 5. PMID 29705387